CLINICAL TRIAL: NCT04477187
Title: Clinical Assessment of Skin Tightening and Contour Change of Submental Tissue Using Bipolar Radiofrequency Microneedling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Jeffrey M. Kenkel, Professor and Chair Department of Plastic Surgery, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU-2020-0593
Record Dates: First submitted 2020-07-08; First posted 2020-07-20 (Actual); Results first posted 2023-12-19 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-11

CONDITIONS: Skin Laxity
MeSH Terms: conditions — Cutis Laxa

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Single Group (Experimental): All subjects will undergo a single treatment for skin laxity in the submentum with a dermal handpiece.
  Interventions: Device: Dermal Handpiece

INTERVENTIONS:
Device: Dermal Handpiece — Radiofrequency (RF) will travel through the RF generator through the electrodes and into the dermal layer beneath the surface of the skin. The microneedles of the dermal cartridges coupled with the thermal heat will stimulate neocollagenesis and neoelastosis, aiding in the reduction of submental laxity.

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of bipolar fractional radiofrequency treatment via use of the Profound System to achieve skin tightening and contour change in lax submental (beneath the chin) tissue.

DETAILED DESCRIPTION:
This is a single-center, unblinded, non-randomized, non-controlled study designed to follow a total of up to 15 qualified and consenting subjects to receive one bipolar fractional radiofrequency microneedling treatment under an IRB approved protocol. Up to 15 subjects will be enrolled and treated at UT Southwestern in the Department of Plastic Surgery. Subjects will be identified from the clinical practice of Dr. Jeffrey Kenkel, Department of Plastic Surgery.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female adults between ages 21-70 years of age.
* Desire skin laxity lift of the submental region.
* Confirmed BMI ≤ 35.
* Subjects who can read, understand, and sign the Informed Consent Form.
* Subjects willing and able to comply with all study requirements.
* Fitzpatrick skin type I-VI.
* Submental fat graded by the Investigator as ≥ 1 using the Clinician-Reported Submental Fat Rating Scale
* Subject is willing not to undergo any type of aesthetic procedure that could confound the study device treatment effects until he/she completes the study.

Exclusion Criteria:

* Active localized or systemic infections, that may alter wound healing.
* Immunocompromised subjects.
* Subjects with coagulation disorder.
* History of skin photosensitivity disorders, or use of photosensitizing drugs (e.g., tetracycline or sulfa drugs).
* Pregnant and/or lactating (All female volunteers will be advised about using birth control during the period of study).
* Excessive skin laxity on the submental and neck (Submental Skin Laxity Grade: SMSLG 4, Appendix E), or other anatomical feature for which reduction in SMF which may, in the judgment of the investigator, result in an aesthetically unacceptable outcome.
* Scarring in areas to be treated.
* Tattoos in the treatment areas to be treated.
* Significant open facial wounds or lesions.
* Severe or cystic acne in treatment areas.
* Current active smoker.
* Use of Accutane (Isotretinoin) within the past 6 months.
* Use of topical retinoids within 48 hours.
* Use of prescription anticoagulants.
* Pacemaker or internal defibrillator.
* History of skin disorders resulting in abnormal wound healing (i.e. keloids, extreme dry and fragile skin).
* Subjects on current oral corticosteroid therapy or within the past 6 months
* Metal implants in the treatment area.
* In the opinion of the investigator, subject is unwilling or unable to adhere to all study requirements, including application and follow-up visits.
* Subjects with a history of radiation therapy to the treatment area.
* Subject has a history of allergy to lidocaine or ester-based local anesthetics.
* Subjects with significant cardiac history or rhythm disturbance who may be unable to tolerate lidocaine with epinephrine.
* Subjects with any skin pathology or condition in the treatment area that could interfere with evaluation or with the use of typical ancillary medical treatments or care used before, during or after treatments (e.g. psoriasis, rosacea, eczema, seborrheic dermatitis, vitiligo, hyper or hypo-skin pigmentation conditions such as post inflammatory hyperpigmentation).
* Subjects who are unwilling to shave excessive hair in the treatment area that might influence or impair evaluation in the opinion of the Investigator.
* Subjects have undergone skin resurfacing or tightening treatments in the treatment area over the past year.
* Subjects have undergone dermatological treatments such as fillers and neurotoxins for the past 6 months in the treatment area.
* Subjects have undergone laser and light treatments in the treatment area over the past 3 months.
* Subjects have undergone superficial peel or microdermabrasion within 4 weeks.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-06-13 (Actual); Study Completion 2022-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Kenkel, MD, Principal Investigator — UT Southwestern
Locations (1):
- UT Southwestern Medical Center- Dept of Plastic Surgery, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Single Group
Started | 15
Completed | 13
Not Completed | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Arm/Group | Single Group
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Fitzpatrick Skin Score [Count of Participants; unit: Participants] — Type I (scores 0-6) always burns, never tans (palest; freckles) Type II (scores 7-13) usually burns, tans minimally (light colored but darker than fair) Type III (scores 14-20) sometimes mild burn, tans uniformly (golden honey or olive)
  Participants
    Skin Type 1 | 2
    Skin Type 2 | 8
    Skin Type 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline of Soft Tissue Surface Area
Description: 3D stereophotogrammetry measurements obtained at Follow Up visits and compared to baseline measurements.
  Percent change from baseline was calculated from baseline for both Month 3 and Month 6.
Time Frame: Month 3 and Month 6 Follow Up
Population: 2 subjects withdrew from the study thus only 13 were analyzed at Month 6.
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- Month 3 Follow Up; 6 Month Follow Up: All subjects will undergo a single treatment for skin laxity in the submentum with a dermal handpiece.
  Dermal Handpiece: Radiofrequency (RF) will travel through the RF generator through the electrodes and into the dermal layer beneath the surface of the skin. The microneedles of the dermal cartridges coupled with the thermal heat will stimulate neocollagenesis and neoelastosis, aiding in the reduction of submental laxity.
Arm/Group | Month 3 Follow Up | 6 Month Follow Up
Number analyzed (Participants) | 15 | 13
percent change | -0.18 (0.89) | -017 (0.32)

2. Primary Outcome: Percent Change From Baseline in Volume
Description: as for outcome 1
Time Frame: Month 3 and Month 6 Follow Up
Population: 2 subjects withdrew from the study thus only 13 were analyzed at Month 6.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Month 3 Follow Up | 6 Month Follow Up
Number analyzed (Participants) | 15 | 13
percent change | -1.30 (0.68) | -1.9 (1.8)

3. Primary Outcome: Percent Change in Minor Tissue Strain
Description: Percent change in Minor Tissue Strain is measured using the Markerless Tracking feature on Canfield's H2 3D Imaging System. 3D stereophotogrammetry measurements obtained at Follow Up visits and compared to baseline measurements.
  Percent change from baseline was calculated from baseline for both Month 3 and Month 6.
Time Frame: Month 3 and Month 6 Follow Up
Population: 2 subjects withdrew from the study thus only 13 were analyzed at Month 6.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Month 3 Follow Up | 6 Month Follow Up
Number analyzed (Participants) | 15 | 13
percentage change | -5.0 (2.5) | -0.44 (0.53)

4. Primary Outcome: Percent Change in Horizontal Displacement
Description: Percent change in Horizontal Displacement is measured using the Markerless Tracking feature on Canfield's H2 3D Imaging System. 3D stereophotogrammetry measurements obtained at Follow Up visits and compared to baseline measurements.
  Percent change from baseline was calculated from baseline for both Month 3 and Month 6.
Time Frame: Month 3 and Month 6 Follow Up
Population: 2 subjects withdrew from the study thus only 13 were analyzed at Month 6.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Month 3 Follow Up | 6 Month Follow Up
Number analyzed (Participants) | 15 | 13
percent change | -0.55 (0.99) | -0.44 (0.53)

5. Primary Outcome: Percent Change in Vertical Displacement
Description: Percent change in Vertical Displacement is measured using the Markerless Tracking feature on Canfield's H2 3D Imaging System. 3D stereophotogrammetry measurements obtained at Follow Up visits and compared to baseline measurements.
  Percent change from baseline was calculated from baseline for both Month 3 and Month 6.
Time Frame: Month 3 and Month 6 Follow Up
Population: 2 subjects withdrew from the study thus only 13 were analyzed at Month 6.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Month 3 Follow Up | 6 Month Follow Up
Number analyzed (Participants) | 15 | 13
percent change | 0.04 (1.06) | -0.19 (0.81)

6. Secondary Outcome: Improvement in Assessments: Global Aesthetic Improvement Score
Description: Blinded reviewers will assessment and score using a 5-point Global Aesthetic Improvement Score (1=Very Much Improved, 5= worse)
Time Frame: Baseline - 6 Months (Day 180)
Population: Only 11 out of 15 enrolled were analyzed since 2 subjects withdrew and the photos of 2 other subjects were not clear.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Blinded Assessment: Clinicians based their evaluation on a comparison of subjects pre- and post- treatment clinical photographs.
Arm/Group | Blinded Assessment
Number analyzed (Participants) | 11
units on a scale | 2.727 (0.49)

7. Secondary Outcome: Subjects Assessment of Pain: Numerical Pain Rating Scale
Description: Immediately after the study procedure, subjects will be asked to rate any pain or discomfort using a 11-point Numerical Pain Rating Scale (0= No pain, 10= Extreme pain)
Time Frame: Visit 2 (Day 0- immediately after study procedure)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Single Group
Number analyzed (Participants) | 13
score on a scale | 1.96 [0.80 to 3.11]

8. Secondary Outcome: Non-invasive Measurements: Transepidermal Water Loss Measurements
Description: Skin texture and laxity will be assessed using non invasive skin measurements.
  Biox Aquaflux- will be used to measure transepidermal water loss.
Time Frame: Baseline, 3 Month and 6 Month Follow Up
Measure: Mean (Standard Deviation); unit: g/m^2/h
Groups:
- Baseline; Month 3 Follow Up; 6 Month Follow Up: All subjects will undergo a single treatment for skin laxity in the submentum with a dermal handpiece.
  Dermal Handpiece: Radiofrequency (RF) will travel through the RF generator through the electrodes and into the dermal layer beneath the surface of the skin. The microneedles of the dermal cartridges coupled with the thermal heat will stimulate neocollagenesis and neoelastosis, aiding in the reduction of submental laxity.
Arm/Group | Baseline | Month 3 Follow Up | 6 Month Follow Up
Number analyzed (Participants) | 15 | 15 | 13
g/m^2/h | 14.084 (3.821) | 11.095 (4.539) | 14.246 (6.661)

9. Secondary Outcome: Non-invasive Measurements: Optical Coherence Tomography (OCT) : [Ra, Rz]
Description: Skin texture and laxity will be assessed using non invasive skin measurements. Skin laxity and elasticity are measured using the Biomechanical Tissue Characterization System.
  Optical coherence tomography (OCT) will be used to topographical and histological images of pre- and post-treated skin.
  Ra, is the average measurement of skin curvatures and takes into all account variances in the skin roughness profile from the center line.
  Rz, is the difference between the highest and lowest data points from the mean surface measurement.
Time Frame: Baseline, 3 months, 6 Months (Day 180)
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Baseline | Month 3 Follow Up | 6 Month Follow Up
Number analyzed (Participants) | 15 | 15 | 13
mm
  Ra (arithmetic mean roughness) | 0.015 (0.004) | 0.014 (0.004) | 0.014 (0.005)
  Rz (Average depth of roughness) | 0.105 (0.027) | 0.1 (0.028) | 0.095 (0.028)

10. Secondary Outcome: Non-invasive Measurements: Optical Coherence Tomography (OCT): Attenuation Coefficient
Description: Skin texture and laxity will be assessed using non invasive skin measurements.
  Optical coherence tomography (OCT) will be used to topographical and histological images of pre- and post-treated skin.
  Attenuation coefficient (AC) is a measure of the decay of light intensity within the sample due to absorption and scattering.
Time Frame: Baseline, 3 months, 6 Months (Day 180)
Measure: Mean (Standard Deviation); unit: mm-1
Arm/Group | Baseline | Month 3 Follow Up | 6 Month Follow Up
Number analyzed (Participants) | 15 | 15 | 13
mm-1 | 4.145 (0.765) | 3.748 (0.674) | 3.661 (0.42)

11. Secondary Outcome: Non-invasive Measurements : Biomechanical Tissue Measurements (Laxity, Elasticity)
Description: Skin laxity and elasticity will be assessed using non invasive skin measurements.
  Bio-Mechanical Tissue Characterization (BTC2000)- will be used to measure skin laxity values of the skin. This is a laser measurement system for objective, quantitative and sensitive analyses of the bio-mechanical properties of: Skin laxity, elasticity.
Time Frame: Baseline, Month 3, Month 6
Measure: Mean (Standard Deviation); unit: mm
Groups:
- Month 3 Follow-up; 6 Month Follow Up: All subjects will undergo a single treatment for skin laxity in the submentum with a dermal handpiece.
  Dermal Handpiece: Radiofrequency (RF) will travel through the RF generator through the electrodes and into the dermal layer beneath the surface of the skin. The microneedles of the dermal cartridges coupled with the thermal heat will stimulate neocollagenesis and neoelastosis, aiding in the reduction of submental laxity.
Arm/Group | Baseline | Month 3 Follow-up | 6 Month Follow Up
Number analyzed (Participants) | 15 | 15 | 13
mm
  Laxity | 1.772 (0.751) | 1.397 (0.624) | 1.197 (0.547)
  Elasticity | 0.997 (0.4) | 1.053 (0.356) | 0.808 (0.387)

12. Secondary Outcome: Non-invasive Measurements : Biomechanical Tissue Measurements (Elastic, Viscoelastic and Ultimate Deformation)
Description: Skin Elastic, Viscoelastic and Ultimate Deformation will be assessed using non invasive skin measurements.
  Bio-Mechanical Tissue Characterization (BTC2000)- will be used to measure skin laxity values of the skin. This is a laser measurement system for objective, quantitative and sensitive analyses of the bio-mechanical properties of: Skin Elastic, Viscoelastic and Ultimate Deformation.
Time Frame: Baseline, Month 3, Month 6
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Baseline | Month 3 Follow-up | 6 Month Follow Up
Number analyzed (Participants) | 15 | 15 | 13
mm
  Elastic Deformation | 3.317 (4.227) | 1.947 (0.591) | 1.718 (0.662)
  Viscoelastic Deformation | 0.098 (0.044) | 0.091 (0.047) | 0.087 (0.043)
  Ultimate Deformation | 2.316 (0.819) | 2.038 (0.621) | 1.805 (0.686)

13. Secondary Outcome: Non-invasive Measurements : Biomechanical Tissue Measurements (Stiffness)
Description: Skin stiffness will be assessed using non invasive skin measurements.
  Bio-Mechanical Tissue Characterization (BTC2000)- will be used to measure skin laxity values of the skin. This is a laser measurement system for objective, quantitative and sensitive analyses of the bio-mechanical properties of: Skin stiffness.
Time Frame: Baseline, Month 3, Month 6
Measure: Mean (Standard Deviation); unit: mmHg/mm
Arm/Group | Baseline | Month 3 Follow-up | 6 Month Follow Up
Number analyzed (Participants) | 15 | 15 | 13
mmHg/mm | 205.129 (50.702) | 208.689 (46.586) | 210.836 (74.519)

14. Secondary Outcome: Non-invasive Measurements : Biomechanical Tissue Measurements (Energy Absorption)
Description: Energy absorption will be assessed using non invasive skin measurements.
  Bio-Mechanical Tissue Characterization (BTC2000)- will be used to measure skin laxity values of the skin. This is a laser measurement system for objective, quantitative and sensitive analyses of the bio-mechanical properties of: Skin - Energy absorption
Time Frame: Baseline, Month 3, Month 6
Measure: Mean (Standard Deviation); unit: mmHg*mm
Arm/Group | Baseline | Month 3 Follow-up | 6 Month Follow Up
Number analyzed (Participants) | 15 | 15 | 13
mmHg*mm | 78.583 (19.482) | 74.724 (21.76) | 76.425 (29.84)

15. Secondary Outcome: Change in Gene Expression at Month 3
Description: Biopsies collected from subjects will be analyzed to observe changes from baseline to Month 3. Gene Expression studies cellular activity and Col1, Col3, ELN, Lox, IL8 are all biomarkers.
  Fold Changes were compared to control and calculated from Ct values of RT-qPCR reactions.
  * Ct: threshold cycle
  * RT-qPCR: Quantitative reverse transcription polymerase chain reaction)
Time Frame: Baseline, Month 3
Population: Inconsistency in the analyzed patients was due to study staff unable to obtain a usable sample during visit.
Measure: Mean (Standard Error); unit: fold change
Groups:
- Month 3: All subjects will undergo a single treatment for skin laxity in the submentum with a dermal handpiece.
  Dermal Handpiece: Radiofrequency (RF) will travel through the RF generator through the electrodes and into the dermal layer beneath the surface of the skin. The microneedles of the dermal cartridges coupled with the thermal heat will stimulate neocollagenesis and neoelastosis, aiding in the reduction of submental laxity.
Arm/Group | Month 3
Number analyzed (Participants) | 7
fold change
  Col1 | 1.18 (0.26)
  Col3 | 1.46 (0.42)
  ELN | 1.27 (0.40)
  Lox | 1.81 (0.39)
  IL8 | 1.81 (5.46)

16. Secondary Outcome: Change in Gene Expression at Month 6
Description: Biopsies collected from subjects will be analyzed to observe changes from baseline to Month 6 . Gene Expression studies cellular activity and Col1, Col3, ELN, Lox, IL8 are all biomarkers.
  Fold Changes were compared to control and calculated from Ct values of RT-qPCR reactions.
  * Ct: threshold cycle
  * RT-qPCR: Quantitative reverse transcription polymerase chain reaction)
Time Frame: Baseline, Month 6
Population: Inconsistency in the analyzed patients was due to study staff unable to obtain a usable sample during visit.
Measure: Mean (Standard Error); unit: fold change
Groups:
- Month 6: All subjects will undergo a single treatment for skin laxity in the submentum with a dermal handpiece.
  Dermal Handpiece: Radiofrequency (RF) will travel through the RF generator through the electrodes and into the dermal layer beneath the surface of the skin. The microneedles of the dermal cartridges coupled with the thermal heat will stimulate neocollagenesis and neoelastosis, aiding in the reduction of submental laxity.
Arm/Group | Month 6
Number analyzed (Participants) | 7
fold change
  Col1 | 6.28 (5.56)
  Col3 | 9.99 (5.56)
  ELN | 2.62 (0.79)
  Lox | 9.24 (8.56)
  IL8 | 9.24 (8.56)

17. Secondary Outcome: Change in Histology at Month 3
Description: All subjects will undergo a single treatment for skin laxity in the submentum with a dermal handpiece.
  Dermal Handpiece: Radiofrequency (RF) will travel through the RF generator through the electrodes and into the dermal layer beneath the surface of the skin. The microneedles of the dermal cartridges coupled with the thermal heat will stimulate neocollagenesis and neoelastosis, aiding in the reduction of submental laxity.
  Fold changes were compared to control and were calculated from fluorescence intensity of a confocal microscopy images.
  Histology studies the structure of the tissue. Col3, Col1, ELN, Macrophage are biomarkers.
Time Frame: Baseline, Month 3
Population: Inconsistency in the analyzed patients was due to study staff unable to obtain a usable sample during visit.
Measure: Mean (Standard Error); unit: fold change
Arm/Group | Month 3 Follow Up
Number analyzed (Participants) | 7
fold change
  Col3 | 1.24 (0.12)
  Col1 | 0.98 (5.77)
  ELN | 1.21 (0.13)
  Macrophage | 0.92 (4.38)

18. Secondary Outcome: Change in Histology at Month 6
Description: All subjects will undergo a single treatment for skin laxity in the submentum with a dermal handpiece.
  Dermal Handpiece: Radiofrequency (RF) will travel through the RF generator through the electrodes and into the dermal layer beneath the surface of the skin. The microneedles of the dermal cartridges coupled with the thermal heat will stimulate neocollagenesis and neoelastosis, aiding in the reduction of submental laxity.
  Histology studies the structure of the tissue. Col3, Col1, ELN, Macrophage are biomarkers.
Time Frame: Baseline, Month 6
Population: Inconsistency in the analyzed patients was due to study staff unable to obtain a usable sample during visit.
Measure: Mean (Standard Error); unit: fold change
Arm/Group | 6 Month Follow Up
Number analyzed (Participants) | 7
fold change
  Col3 | 1.04 (0.16)
  Col1 | 0.93 (5.04)
  ELN | 0.98 (0.18)
  Macrophage | 0.89 (5.55)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Single Group
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-18): https://cdn.clinicaltrials.gov/large-docs/87/NCT04477187/Prot_SAP_002.pdf